CLINICAL TRIAL: NCT03185429
Title: Study of DC Vaccine Loaded Tumor Specific Antigen in Treating Patients With Gastrointestinal Solid Tumor
Brief Title: TSA-DC Vaccine in Treating Patients With Gastrointestinal Solid Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BGI, China (Other)
Collaborators: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGI-002
Record Dates: First submitted 2017-06-11; First posted 2017-06-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Tumor Gastric; Tumor, Colorectal
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Drug:Cyclophosphamide
  Biological/Vaccine:Tumor Specific Antigen-loaded Dendritic Cells
  Interventions: Biological: Tumor Specific Antigen-loaded Dendritic Cells; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Tumor Specific Antigen-loaded Dendritic Cells — Subjects will be given subcutaneous injection of 5.0x10^6-1.0x10^7 TSA-DC on week 1,3,5,11,17,23,35,47.
  Other Names: TSA-DC vaccine
Drug: Cyclophosphamide — 300 mg/m2 by vein before the first cell infusion.
  Other Names: Cytoxan

SUMMARY:
The goal of this study is to learn about the safety and tolerance of autologous TSA-DC cell and evaluate the efficacy and feasibility of the cell therapy compared to the patients' past standard regimen. 20 gastrointestinal solid tumors subjects failed from at least one systemic therapy will be enrolled into the trial and receive a succession of treatment of TSA-DC vaccine.

DETAILED DESCRIPTION:
20 gastrointestinal solid tumor subjects failed from at least one systemic therapy will be enrolled into the trial .Subjects will be given subcutaneous injection of 5.0x10^6-1.0x10^7 TSA-DC on week 1, 3, 5, 11,17,23,35,47. Before the first cell infusion, the subjects should undergo a non-myeloablative chemotherapy regimen of Cyclophosphamide 300mg/m2 iv. Radiologic tumor assessment will be repeated every 8 weeks during treatment, until time of progression. Treatment will continue until disease progression, intolerance of toxic , withdrawal from the study, study completion, or study termination.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 and ≤75,no gender based;
2. Expression of HLA-A0201/1101/2402;
3. Histopathologic documentation of gastrointestinal solid tumors(stomach cancer or colorectal cancer ) concurrent with the diagnosis of metastatic disease, and the tumor is Measurable;
4. Patients must have adequate tissue (fresh or paraffin block) for DNA extraction, which is used for gene sequencing, and prognoses the tumor specific antigen in turn,can predict to have new tumor antigens with high affinity for MHC molecules;
5. Failure in conventional treatment， or though benefit from chemotherapy the patient can't tolerant subjectively;
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2 and an anticipate life expectancy of at least three months,be cooperate to adverse reactions monitoring and therapeutic evaluation of the treatment;
7. Participants of child-bearing potential must agree to use adequate contraceptive methods up to 12 months after the pretreatment;
8. Serology：Seronegative for HIV antibody,seronegative for hepatitis C antibody. Hematology：Absolute neutrophil count ≥ 1000/mm(3) without the support of filgrastim ,WBC ≥ 3000/mm(3)，lymphocyte count ≥ 800/mm(3)，Platelet count ≥ 100,000/mm(3)，Hemoglobin ≥ 9.0 g/dl Chemistry：Serum ALT/AST ≤ 2.5 times the upper limit of normal，Serum Creatinine ≤1.6 mg/dl，Total bilirubin < 1.5 mg/dl, except in patients with Gilbert s Syndrome who must have a total bilirubin < 3.0 mg/dl;
9. Patients or their legal representatives are willing and able to understand and written informed consent form for the trial;

Exclusion Criteria:

1. Is pregnant or breastfeeding,or expecting to conceive;
2. Have a history of severe immediate hypersensitivity reaction to any of the agents used in this study.
3. Suffered grade 3-4 major organ immune-related adverse events after anti-PD1/PDL1 antibody treatment.
4. Once received allogeneic organ transplantation (including bone marrow transplantation and peripheral stem cell transplantation, except for corneal transplantation);
5. Have clinical symptoms of central nervous system metastases;
6. Have used a large number of glucocorticoids or other immunosuppressive agents within 4 weeks;
7. Have any active autoimmune disease ;
8. Be in active infection or undergo an unknown cause fever> 38.5 ℃ during screening or before the first administration(except tumor fever which evaluated by the researchers have no effect to enrollment );
9. Received chemotherapy or small molecule targeted drug therapy in 4 weeks prior to chemotherapy pretreatment;
10. Received any antibody drug therapy (including PD-1 and CTLA-4) within 6 weeks before the treatment period;
11. Severe liver and kidney dysfunction or uncontrollable diabetes, hypertension and other chronic systemic diseases; severe coagulation disorders, mental illness, cardiopulmonary disease，hydrothorax or ascites;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
safety endpoint | one year
  All the local or systemic reactions, adverse events and serious adverse events that occurred between the first and the second TSA-DC administration.
Overall Response Rate | one year
  Percentage of cases whose tumor shrinks to a certain extent and remains for a certain period of time.
Proportion of the number of cases that has produced tumor-specific antigen-specific T cells in peripheral blood. | one year

SECONDARY OUTCOMES:
Secondary safety endpoint | one year
  All local or systemic reactions, adverse events and serious adverse events that occurred from entering the trial until 30 days after the last treatment;
Six month DCR(CRR+PRR+SDR) | 6 month
  Percentage of cases with no progression (CR + PR + SD) in 6 months after initiation of treatment;
Duration of Response(DOR) | one year
  The time from the first tumor evaluation of remission(CR + PR ) till the first assessment of PD or the end the study.
Progression-free survival(PFS) | one year
  The time from entering the trial till the subject has been diagnosed with progression of disease or died.
rate of 12-month survival | one year
  Percentage of cases with 12 months survival after initiation of treatment in all the subjects;
Quality score of life improvement | one year
  Evaluated by the questionnaire of life improvement quality collected from the screening to treatment periods.

CONTACTS AND LOCATIONS:
Overall Officials: ZengQing Guo, Professor, Principal Investigator — Fujian Cancer Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chiang CL, Kandalaft LE, Tanyi J, Hagemann AR, Motz GT, Svoronos N, Montone K, Mantia-Smaldone GM, Smith L, Nisenbaum HL, Levine BL, Kalos M, Czerniecki BJ, Torigian DA, Powell DJ Jr, Mick R, Coukos G. A dendritic cell vaccine pulsed with autologous hypochlorous acid-oxidized ovarian cancer lysate primes effective broad antitumor immunity: from bench to bedside. Clin Cancer Res. 2013 Sep 1;19(17):4801-15. doi: 10.1158/1078-0432.CCR-13-1185. Epub 2013 Jul 9. PMID 23838316
- [Background] Schuler PJ, Harasymczuk M, Visus C, Deleo A, Trivedi S, Lei Y, Argiris A, Gooding W, Butterfield LH, Whiteside TL, Ferris RL. Phase I dendritic cell p53 peptide vaccine for head and neck cancer. Clin Cancer Res. 2014 May 1;20(9):2433-44. doi: 10.1158/1078-0432.CCR-13-2617. Epub 2014 Feb 28. PMID 24583792
- [Background] Carreno BM, Magrini V, Becker-Hapak M, Kaabinejadian S, Hundal J, Petti AA, Ly A, Lie WR, Hildebrand WH, Mardis ER, Linette GP. Cancer immunotherapy. A dendritic cell vaccine increases the breadth and diversity of melanoma neoantigen-specific T cells. Science. 2015 May 15;348(6236):803-8. doi: 10.1126/science.aaa3828. Epub 2015 Apr 2. PMID 25837513